CLINICAL TRIAL: NCT03000777
Title: An Unicentric, Double-blind, Placebo Controlled, Phase IV Clinical Trial of Oral Melatonin Plus Zinc to Evaluate Relieving Self-reported Fatigue in CFS/ME
Brief Title: Oral Melatonin Plus Zinc Supplementation in Chronic Fatigue Syndrome/Myalgic Encephalomyelitis (CFS/ME)
Acronym: MELATOZINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Viñas, S.A. (Industry)
Collaborators: Hospital Vall d'Hebron (Other); Laboratorio Echevarne (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC/LV/MEL-ZN/SFC
Record Dates: First submitted 2016-12-19; First posted 2016-12-22 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Fatigue Syndrome, Chronic; Myalgic Encephalomyelitis
Keywords: melatonin; zinc; Myalgic Encephalomyelitis; Chronic Fatigue Syndrome; sleep; pain
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Pain | interventions — Melatonin; Zinc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin plus Zinc (Experimental): Melatonin plus Zinc
  Interventions: Dietary Supplement: melatonin plus zinc
- Placebo (Placebo Comparator): Isomaltose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: melatonin plus zinc — Melatonin 1 mg plus Zinc 10 mg o.d. 1 hour before going to bed during 16 weeks
  Other Names: MelatoZinc
  Arms: Melatonin plus Zinc
Other: Placebo — Isomaltose o.d. 1 hour before going to bed during 16 weeks
  Other Names: Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of oral melatonin plus zinc supplementation in relieving self-reported fatigue in CFS/ME

DETAILED DESCRIPTION:
Chronic Fatigue Syndrome/Myalgic Encephalomyelitis (CFS/ME) is a complex medical condition, characterized by severe disabling fatigue with no known cause, no established diagnostic tests, and no universally effective treatment. No studies have evaluated symptomatic treatment using oral melatonin plus zinc supplementation in CFS/ME. The primary endpoint was to assess the effect of melatonin plus zinc supplementation on self-reported fatigue. Secondary measures included self-reported outcomes of sleep problems, anxiety/depression, dysautonomia, QoL and side-effects during treatment.

ELIGIBILITY:
Inclusion Criteria:

* CFS patient based on the 1994 Centers for Disease Control and Prevention/Fukuda definition.
* Patient who provided signed informed consent.

Exclusion Criteria:

* Patients who are participating in another clinical trial of the same or different nature previous 30 days prior to inclusion.
* Any subject that, in the judgment of the investigator, is not able to follow the instructions or to perform a good completion of the treatment.
* Subjects that do not provide signed informed consent.
* Patients who are receiving any of the drugs or products that may interfere with the results, and whose withdrawal could be a relevant medical problem.
* Patients receiving oral anticoagulants.
* Pregnancy or lactation
* Patients with hypersensitivity to melatonin and/or zinc.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
To evaluate relieving self-reported fatigue using the Fatigue Impact Scale 40-items (FIS 40) questionnaire after oral melatonin plus zinc administration | within the first 16 weeks (plus 4 weeks with no treatment)

SECONDARY OUTCOMES:
Side effects during treatment. | within the first 16 weeks (plus 4 weeks with no treatment)
Self-reported sleep quality through the Pittsburgh Sleep Quality Index (PSQI) questionnaire. | within the first 16 weeks (plus 4 weeks with no treatment)
Self-reported anxiety/depression through the Hospital Anxiety and Depression Scale (HADS) questionnaire. | within the first 16 weeks (plus 4 weeks with no treatment)
Self-reported dysautonomia using the Composite Autonomic Symptom Score 31-items (COMPASS 31) questionnaire. | within the first 16 weeks (plus 4 weeks with no treatment)
Self-reported QoL through the Short Form Health Survey 36-items (SF-36) questionnaire. | within the first 16 weeks (plus 4 weeks with no treatment)

CONTACTS AND LOCATIONS:
Overall Officials: José Alegre, MD; PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro-Marrero J, Cordero MD, Saez-Francas N, Jimenez-Gutierrez C, Aguilar-Montilla FJ, Aliste L, Alegre-Martin J. Could mitochondrial dysfunction be a differentiating marker between chronic fatigue syndrome and fibromyalgia? Antioxid Redox Signal. 2013 Nov 20;19(15):1855-60. doi: 10.1089/ars.2013.5346. Epub 2013 May 29. PMID 23600892
- [Background] Castro-Marrero J, Cordero MD, Segundo MJ, Saez-Francas N, Calvo N, Roman-Malo L, Aliste L, Fernandez de Sevilla T, Alegre J. Does oral coenzyme Q10 plus NADH supplementation improve fatigue and biochemical parameters in chronic fatigue syndrome? Antioxid Redox Signal. 2015 Mar 10;22(8):679-85. doi: 10.1089/ars.2014.6181. Epub 2014 Dec 18. PMID 25386668
- [Background] Castro-Marrero J, Saez-Francas N, Segundo MJ, Calvo N, Faro M, Aliste L, Fernandez de Sevilla T, Alegre J. Effect of coenzyme Q10 plus nicotinamide adenine dinucleotide supplementation on maximum heart rate after exercise testing in chronic fatigue syndrome - A randomized, controlled, double-blind trial. Clin Nutr. 2016 Aug;35(4):826-34. doi: 10.1016/j.clnu.2015.07.010. Epub 2015 Jul 17. PMID 26212172
- [Background] Saez-Francas N, Calvo N, Alegre J, Castro-Marrero J, Ramirez N, Hernandez-Vara J, Casas M. Childhood trauma in Chronic Fatigue Syndrome: focus on personality disorders and psychopathology. Compr Psychiatry. 2015 Oct;62:13-9. doi: 10.1016/j.comppsych.2015.06.010. Epub 2015 Jun 17. PMID 26343462
- [Background] Faro M, Saez-Francas N, Castro-Marrero J, Aliste L, Fernandez de Sevilla T, Alegre J. Gender differences in chronic fatigue syndrome. Reumatol Clin. 2016 Mar-Apr;12(2):72-7. doi: 10.1016/j.reuma.2015.05.007. Epub 2015 Jul 17. English, Spanish. PMID 26190206
- [Background] Calvo N, Saez-Francas N, Valero S, Alegre J, Casas M. Comorbid personality disorders in chronic fatigue syndrome patients: a marker of psychopathological severity. Actas Esp Psiquiatr. 2015 Mar-Apr;43(2):58-65. Epub 2015 Mar 1. PMID 25812543
- [Background] Faro M, Alegre J. [Fibromyalgia as a comorbid phenomenon in autoinflammatory diseases]. Med Clin (Barc). 2015 Jun 8;144(11):525. doi: 10.1016/j.medcli.2014.07.033. Epub 2014 Nov 26. No abstract available. Spanish. PMID 25433788
- [Background] Santamarina-Perez P, Eiroa-Orosa FJ, Rodriguez-Urrutia A, Qureshi A, Alegre J. Neuropsychological impairment in female patients with chronic fatigue syndrome: a preliminary study. Appl Neuropsychol Adult. 2014;21(2):120-7. doi: 10.1080/09084282.2013.771264. Epub 2013 Aug 13. PMID 24826505
- [Background] Saez-Francas N, Valero S, Calvo N, Goma-I-Freixanet M, Alegre J, de Sevilla TF, Casas M. Chronic fatigue syndrome and personality: a case-control study using the Alternative Five Factor Model. Psychiatry Res. 2014 May 30;216(3):373-8. doi: 10.1016/j.psychres.2014.02.031. Epub 2014 Mar 3. PMID 24630915
- [Background] Docampo E, Escaramis G, Gratacos M, Villatoro S, Puig A, Kogevinas M, Collado A, Carbonell J, Rivera J, Vidal J, Alegre J, Estivill X, Rabionet R. Genome-wide analysis of single nucleotide polymorphisms and copy number variants in fibromyalgia suggest a role for the central nervous system. Pain. 2014 Jun;155(6):1102-1109. doi: 10.1016/j.pain.2014.02.016. Epub 2014 Feb 26. PMID 24582949
- [Background] Faro M, Saez-Francas N, Castro-Marrero J, Aliste L, Collado A, Alegre J. [Impact of the fibromyalgia in the chronic fatigue syndrome]. Med Clin (Barc). 2014 Jun 16;142(12):519-25. doi: 10.1016/j.medcli.2013.06.030. Epub 2014 Jan 2. Spanish. PMID 24387955
- [Background] Blazquez A, Ruiz E, Aliste L, Garcia-Quintana A, Alegre J. The effect of fatigue and fibromyalgia on sexual dysfunction in women with chronic fatigue syndrome. J Sex Marital Ther. 2015;41(1):1-10. doi: 10.1080/0092623X.2013.864370. Epub 2014 Mar 11. PMID 24274008
- [Background] Valero S, Saez-Francas N, Calvo N, Alegre J, Casas M. The role of neuroticism, perfectionism and depression in chronic fatigue syndrome. A structural equation modeling approach. Compr Psychiatry. 2013 Oct;54(7):1061-7. doi: 10.1016/j.comppsych.2013.04.015. Epub 2013 Jun 5. PMID 23759150
- [Background] Curriu M, Carrillo J, Massanella M, Rigau J, Alegre J, Puig J, Garcia-Quintana AM, Castro-Marrero J, Negredo E, Clotet B, Cabrera C, Blanco J. Screening NK-, B- and T-cell phenotype and function in patients suffering from Chronic Fatigue Syndrome. J Transl Med. 2013 Mar 20;11:68. doi: 10.1186/1479-5876-11-68. PMID 23514202
- [Derived] Castro-Marrero J, Zaragoza MC, Lopez-Vilchez I, Galmes JL, Cordobilla B, Maurel S, Domingo JC, Alegre-Martin J. Effect of Melatonin Plus Zinc Supplementation on Fatigue Perception in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: A Randomized, Double-Blind, Placebo-Controlled Trial. Antioxidants (Basel). 2021 Jun 23;10(7):1010. doi: 10.3390/antiox10071010. PMID 34201806